CLINICAL TRIAL: NCT05838638
Title: Serious Gaming for Chemotherapy-induced Nausea and Vomiting in Older Adults With Cancer: A Randomized Clinical Trial
Brief Title: Serious Gaming for Chemotherapy-induced Nausea and Vomiting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Orlando Health, Inc. (Other); University of Miami (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003808; R01NR020003 (NIH)
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Chemotherapy-induced Nausea and Vomiting
Keywords: aged; digital technology; nausea; neoplasm; Drug related side effects and adverse reactions; self-management
MeSH Terms: conditions — Neoplasms; Vomiting; Nausea; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This intervention is a serious game which allows older adults under treatment for cancer to practice making self-care decisions for an avatar that is being sent home after their first chemotherapy treatment. This serious game is coupled with a discussion with the research assistant about choices related to managing nausea and vomiting at home
  Interventions: Behavioral: eSSET-CINV
- Control (Active Comparator): The control group will receive standard education related to managing nausea and vomiting and will have the opportunity to participate in the intervention at the end of the study
  Interventions: Behavioral: eSSET-CINV

INTERVENTIONS:
Behavioral: eSSET-CINV — Participants in the intervention group will be asked to play the serious game on an iPad at their first chemotherapy treatment visit. The control group will be able to play at time 6.
  Other Names: Managing at Home- CINV

SUMMARY:
The purpose of this study is to examine the effectiveness of a technology-based intervention for managing nausea and vomiting in older adults with cancer. Participants will be randomized to either an intervention or control group. Outcomes such as symptom severity, quality of life, and resource use will be examined.

DETAILED DESCRIPTION:
The goal of this study is to increase the use of preventative self-management behaviors for nausea and vomiting in older adults receiving chemotherapy to reduce negative outcomes and emergency or hospital admissions. Early reinforcement of standard education and re-framing any preconceived beliefs about the ability of nausea and vomiting to be managed will increase preventative self-management behaviors and improve patient outcomes. Participants will be in the study for 6 chemotherapy treatment cycles. This could be 12 to 24 weeks depending on if they receive treatment every 2, 3 or 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 60 or older
* newly diagnosed with cancer
* treatment with any chemotherapeutic agent of moderate or high emetic potential
* on a 2, 3 or 4 week treatment cycle
* proficient in English
* has a telephone

Exclusion Criteria:

* previous diagnosis and/or treatment for cancer
* end stage disease with less than 6 months to live
* visually or hearing impaired without corrective device

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Healthcare resource use | From baseline through the end of the study at 12 or 24 weeks
  any emergency department or hospital admission will be recorded using a dichotomous variable (yes/no)
CINV severity | From baseline1 through the end of the study at 12 or 24 weeks
  The Symptom Management Checklist will measure the presence and severity of nausea and vomiting. Participants will be sent a text link every day for 6 days after chemotherapy or complete this data on a form at home. This starts right after time 1. Nausea will be reported on a 0-10 scale. Higher numbers equal more nausea.

SECONDARY OUTCOMES:
Self-management behaviors | From baseline through the end of the study at 12 or 24 weeks
  The Symptom Management Checklist will measure self-management behaviors and preventive behaviors for CINV. Participants will be sent a text link every day for 6 days after chemotherapy or complete this data on a form at home. This starts right after Time 1.
Symptom severity | Baseline and 12 or 24 weeks
  The Symptom Representation Questionnaire Part 1 is a 24 item self-report measure that will be used to identify the presence and severity of common treatment-related side effects (0 to 10 scale). Higher numbers indicate more severe symptoms. This measure asks participants to think about their symptoms over the last week
Cognitive representation | Baseline and 12 or 24 weeks
  The Symptom Representation Questionnaire Part 2 has 15 questions related to cognitive beliefs about nausea. Sub scales examine symptom cause, timeline, cure/control, and consequences. An agreement type Likert scale is used.
Health-related Quality of Life | baseline, 4,8,12,16,20, and 24 weeks
  The EORTC-30 will measure quality of life at each treatment cycle. Higher scores mean better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Loerzel, PhD, Principal Investigator — University of Central Florida
Locations (2):
- United States (2):
  - Miller School of Medicine Sylvester Comp. Cancer Center, Miami, Florida
  - Orlando Health, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loerzel V. Cognitive Representation of Treatment-Related Symptoms in Older Adults With Cancer. Cancer Nurs. 2017 May/Jun;40(3):230-236. doi: 10.1097/NCC.0000000000000395. PMID 27271365
- [Background] Loerzel V, Clochesy J, Geddie P. Using a community advisory board to develop a serious game for older adults undergoing treatment for cancer. Appl Nurs Res. 2018 Feb;39:207-210. doi: 10.1016/j.apnr.2017.11.030. Epub 2017 Nov 21. PMID 29422160
- [Background] Loerzel VW, Hines RB, Deatrick CW, Geddie PI, Clochesy JM. Unplanned emergency department visits and hospital admissions of older adults under treatment for cancer in the ambulatory/community setting. Support Care Cancer. 2021 Dec;29(12):7525-7533. doi: 10.1007/s00520-021-06338-y. Epub 2021 Jun 9. PMID 34105026
- [Background] Wochna Loerzel V, Clochesy JM, Geddie PI. Using Serious Games to Increase Prevention and Self-Management of Chemotherapy-Induced Nausea and Vomiting in Older Adults With Cancer. Oncol Nurs Forum. 2020 Sep 1;47(5):567-576. doi: 10.1188/20.ONF.567-576. PMID 32830802
- [Derived] Loerzel V, Alamian A, Clochesy J, Geddie PI. Serious Gaming for Chemotherapy-Induced Nausea and Vomiting in Older Adults With Cancer: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2024 Oct 2;13:e64673. doi: 10.2196/64673. PMID 39357051